CLINICAL TRIAL: NCT06887907
Title: Phenotypic and Transcriptomic Description of Megakaryocytes in Sickle Cell Patient
Acronym: MEGADREP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/25/0017
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: Megakaryocyte; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample withdraw from sickle cell disease patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Sickle cell disease patients at rest since at least 1 year: Patient at steady state since at least 1 year
- Sickle cell disease patients at rest: Patient at steady state (without crises)
- Vaso-occlusive crisis: Sickle cell disease patients during vaso-occlusive crisis
- Acute chest syndrome: Sickle cell disease patients during acute chest syndrome

SUMMARY:
Sickle cell disease is the most common inherited blood disorder in the world. Chronic hemolysis induces platelet activation and chronic inflammation. Platelets and megakaryocyte, as medullar platelets precursors, are known to play a role in innate immunity. Little is known about the role of megakaryocytes at basal state and during acute complication in sickle cell disease patients. The aim of this study is to evaluate the role of megakaryocytes in sickle cell disease.

DETAILED DESCRIPTION:
Sickle cell disease is the most common inherited blood disorder worldwide. It is a hemoglobinopathy characterized by a chronic hemolysis, vaso-occlusion, endotheliopathy, coagulation activation and chronic inflammation. It is a multisystemic disease leading to acute (Vaso-occlusive crisis, acute chest syndrome) and chronic complications with multiorgan damage. Platelets are activated and release pro-inflammatory mediators in sickle cell disease patients. Less is known about megakaryocytes, precursors of platelets, in sickle cell disease. Nevertheless, it recently has been shown that megakaryocytes, are also produced in the lung and can displayed a pro-inflammatory transcriptomic signature depending on local conditions. An increase in pulmonary megakaryocytes has been described in vascular diseases associated with excessive coagulation, in acute respiratory distress syndrome, and infections demonstrated that during severe SARS-CoV2 pneumonia, there was an increase in circulating megakaryocytes characterized by a pro-inflammatory transcriptomic signature. Acute chest syndrome represents the first cause of mortality in patients with sickle cell disease, characterized by an acute respiratory failure whose pathophysiology includes vaso-occlusive phenomena, infection and inflammation. Given a pro-inflammatory and pro-thrombotic state in sickle cell disease, particularly in acute chest syndrome, we suggest that the megakaryocyte may be involved in the pathophysiology of sickle cell disease. The aim of this study is to evaluate the role of megakaryocytes by peripheral blood sampling from 10 sickle cell disease patients at rest since at least 1 year, 10 sickle cell disease patients at rest and 20 patients during acute complications (10 sickle cell disease patients during vaso-occlusive crises, 10 sickle cell disease patients during acute chest syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease SS or S-béta° thalassemia
* Patient at steady state since at least 1 year or at steady state (without crisis), or during vaso-occlusive crisis or during acute chest syndrome
* Age > 18 years old

Exclusion Criteria:

* Patient objects to take part in the study Hematologic disorder (leukemia, myeloma, myelodysplasic syndrome, myeloproliferative syndrome)
* Immune thrombocytopenia, Immunosuppressive or anti-inflammatory (biotherapies, corticosteroids, non steroidal anti-inflammatories drugs) Page 12 sur 23
* Anti-platelets agents
* Red blood cell exchange or transfusion < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient from CHU de Toulouse at steady state since at least 1 year or at steady state (without crisis), or during vaso-occlusive crisis or during acute chest syndrome
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Description of circulant megakaryocytes | 12 months
  Phenotypic and transcriptomic description of circulant megakaryocytes in sickle cell patient

CONTACTS AND LOCATIONS:
Overall Officials: Pierre COUGOUL, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France, France